CLINICAL TRIAL: NCT06614179
Title: A Pan-cancer Screening and Diagnosis Model Based on Abdominal CT Was Established
Status: Recruiting | Type: Observational
Sponsor: Xiangdong Cheng (Other)
Responsible Party: Sponsor-Investigator, Xiangdong Cheng, Professor, Zhejiang Cancer Hospital
Organization: Zhejiang Cancer Hospital (Other)
Other Study IDs: IIT-2024-279
Record Dates: First submitted 2024-09-01; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Abdominal Neoplasm
MeSH Terms: conditions — Abdominal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Abdominal noncontrast scan and contrast-enhanced CT were used to establish a screening and diagnostic model for abdominal tumors

DETAILED DESCRIPTION:
Secondary objective: To establish a grading model of abdominal tumors based on clinical indicators Exploratory Objective: To include CT scans in large-scale non-tumor populations for validation and to improve model accuracy Certainty

ELIGIBILITY:
Inclusion Criteria:

* Patients with abdominal tumors:
* all patients were pathologically diagnosed with abdominal tumors;
* The clinical case data of all patients were complete, and complete follow-up was obtained, with clear information on medical visits, operation time and survival status within 2 years. If the cause of death is unknown, it will be recorded as censored data;
* All patients had no history of active abdominal bleeding, no serious infection or other abdominal diseases that affected the observation of CT imaging within 3 months before surgery.
* Non-tumor population:
* all patients have complete clinical case data, complete abdominal CT, no history of malignant tumors, no serious infections or other abdominal diseases that affect the diagnosis and observation of CT imaging.

Exclusion Criteria:

* Cases in which contrast-enhanced or noncontrast CT images show unclear lesions, with significant noise and artifacts;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with abdominal tumors or Non-tumor population
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Whether or not there is a diagnosis of abdominal tumor questionnaire | first visited at baseline
  Whether or not there is a diagnosis of abdominal tumor

CONTACTS AND LOCATIONS:
Overall Officials: Xiangdong Cheng, Principal Investigator — Zhejiang Cancer Hospital
Locations (2):
- China (2):
  - Cancer Hospital of the University of Chinese Academy of Sciences (Zhejiang Cancer Hospital), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital；Cancer hospital of the university of chinese academy of sciences, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Abdominal noncontrast scan and contrast-enhanced CT were used to establish a screening and diagnostic model for abdominal tumors
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Hu C, Xia Y, Zheng Z, Cao M, Zheng G, Chen S, Sun J, Chen W, Zheng Q, Pan S, Zhang Y, Chen J, Yu P, Xu J, Xu J, Qiu Z, Lin T, Yun B, Yao J, Guo W, Gao C, Kong X, Chen K, Wen Z, Zhu G, Qiao J, Pan Y, Li H, Gong X, Ye Z, Ao W, Zhang L, Yan X, Tong Y, Yang X, Zheng X, Fan S, Cao J, Yan C, Xie K, Zhang S, Wang Y, Zheng L, Wu Y, Ge Z, Tian X, Zhang X, Wang Y, Zhang R, Wei Y, Zhu W, Zhang J, Qiu H, Su M, Shi L, Xu Z, Zhang L, Cheng X. AI-based large-scale screening of gastric cancer from noncontrast CT imaging. Nat Med. 2025 Sep;31(9):3011-3019. doi: 10.1038/s41591-025-03785-6. Epub 2025 Jun 24. PMID 40555751